CLINICAL TRIAL: NCT05407051
Title: Investigating Effects of Family-Centered Treatment for Depression in Primary Care for Hispanic Youth
Brief Title: Family-Centered Treatment for Depression in Hispanic Youth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000028
Record Dates: First submitted 2022-05-25; First posted 2022-06-07 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Depression; Family Research; Teen Depression
Keywords: teen depression; hispanic; family centered
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): In the Treatment as Usual condition, parents will simply be given a list of mental health referrals and crisis numbers.
  Interventions: Behavioral: Treatment as Usual
- Family Centered Treatment (Experimental): In the Family-Centered Treatment Arm, parents would be given the same list of mental health referrals and crisis numbers, but in this condition, they would authorize researchers to share their contact information with the partner agency, Catholic Charities, and would then be linked directly to bilingual adult mental health services there with a behavioral health provider who would provide collateral therapy to parents via telehealth. Although parents will be referred to the community partner for therapy as a part of the research intervention, the behavioral health providers at the community partner will be providing therapy as they usually do for these participants in line with their usual job duties.
  Interventions: Behavioral: Family Centered Treatment

INTERVENTIONS:
Behavioral: Family Centered Treatment — In the Family-Centered Treatment Arm, parents would be given the same list of mental health referrals and crisis numbers, but in this condition, they would authorize researchers to share their contact information with the partner agency, Catholic Charities, and would then be linked directly to bilingual adult mental health services there with a behavioral health provider who would provide collateral therapy to parents via telehealth. Although parents will be referred to the community partner for therapy as a part of the research intervention, the behavioral health providers at the community partner will be providing therapy as they usually do for these participants in line with their usual job duties.
  Arms: Family Centered Treatment
Behavioral: Treatment as Usual — All participants (parents) would receive follow-up calls from a MetroHealth research personnel at 3 months and 6 months to measure changes in parent mental health outcomes, as well as satisfaction.
  Children of parents in both conditions will receive treatment as usual which includes brief consultation for 3-5 sessions with an integrated MetroHealth behavioral health provider which is already standard practice in the clinic. Sessions typically occur monthly. Teens will be re-administered the Patient Health Questionnaire -9 by the integrated behavioral health provider as a part of clinical practice to measure treatment progress and this information will be obtained at the end of 6 months of treatment via chart review (see data sheet). Repeated measurement of patient's symptoms over the course of several months of treatment is common in clinical practice to measure patient's symptom improvement.
  Arms: Treatment as Usual

SUMMARY:
Studies suggest that for youth in poverty, addressing stressors like parental mental health concerns may improve children's mental health outcomes. Rates of depression and suicidality are growing among teens nationwide and rates of depression are disproportionately high for Hispanic youth. Hispanic families are disproportionately impacted by poverty and are disproportionately exposed to adverse childhood experiences, yet Hispanic patients are less likely than non-Hispanic patient to have access to specialty mental healthcare. Integrating mental health care into primary care is one avenue towards making specialized mental healthcare more accessible to the Hispanic community. There have been few studies focused on addressing parental mental health within pediatric primary care, and even fewer focused specifically on supporting Hispanic families within primary care. The current study would seek to formally assess whether a family-centered treatment approach improves depression outcomes for both Hispanic teens and parents identified in primary care.

The current study would implement depression screening for teens and global mental health screening for parents in MetroHealth's Pediatric Hispanic Clinic. Teens identified with depression would receive integrated consultation with a psychology provider as usual. In this study, parents who agree to participate would also be screened for depression, anxiety, trauma and parenting stress. Parents who screen positive would then be randomized to receive either a list of referrals for bilingual mental health services in the community (treatment as usual), or into the family-centered treatment arm. In the family-centered treatment arm, parents would be connected directly to bilingual adult mental health services with a community partner, Catholic Charities, who would provide collateral therapy to parents via telehealth. Families will then receive follow-up calls from a bilingual MetroHealth provider 3- and 6-months later to re-administer the same parent outcome measures.

Investigators hypothesize that adolescent depression symptoms will improve to a greater degree in the family-centered treatment condition as compared to treatment as usual, and that measures of parental mental health and parenting stress will show significantly greater improvement in the family-centered treatment condition as compared to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Teens 12+ seen in pediatric Hispanic clinic will be screened using the Patient Health Questionnaire -9 for depression as a part of standard clinic protocols. Parents of teens 12+ who screen positive for depression who also screen positive for mental health concerns may be included in the study. Parents who participate in the initial survey but who do NOT screen positive for any of their own mental health concerns will be given a list of mental health referrals and crisis numbers but will not be eligible to participate in the rest of the study or any follow-up calls.

Parents or legal guardians may be included in the study if their teen is over the age of 12, being seen in the pediatric Hispanic clinic, screens positive for depression during pediatric visit, and if parents then screen positive for any mental health concern during the initial survey.

Exclusion Criteria:

* Adults unable to consent
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 | baseline, 3 and 6 month change
  Measure of Depression - score ranges from 0-27 with higher scores indicating more symptoms of depression
Change in Generalized Anxiety Disorder-7 | baseline, 3 and 6 month change
  Measure of Anxiety - score range from 0-21 with higher score indicating more symptoms of anxiety

SECONDARY OUTCOMES:
Change in Post Traumatic Stress Disorder CheckList - for Civilians | baseline, 3 and 6 month change
  Measure of Post Traumatic Stress disorder -score ranges from 17-85 with higher scores indicating more symptoms of Post Traumatic Stress
Change in Parenting Stress Index -4 | baseline, 3 and 6 month change
  Parenting stress index - raw scores are calculated and converted to percentiles with specified cutoffs for each subscale. Higher percentiles indicate higher levels of parenting stress.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Myers, PhD, Principal Investigator — MetroHealth Systems
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slopen N, Fitzmaurice G, Williams DR, Gilman SE. Poverty, food insecurity, and the behavior for childhood internalizing and externalizing disorders. J Am Acad Child Adolesc Psychiatry. 2010 May;49(5):444-52. doi: 10.1097/00004583-201005000-00005. PMID 20431464
- [Background] Friedman SH, McEwan MV. Treated Mental Illness and the Risk of Child Abuse Perpetration. Psychiatr Serv. 2018 Feb 1;69(2):211-216. doi: 10.1176/appi.ps.201700120. Epub 2017 Nov 1. PMID 29089007
- [Background] Pilowsky DJ, Wickramaratne P, Talati A, Tang M, Hughes CW, Garber J, Malloy E, King C, Cerda G, Sood AB, Alpert JE, Trivedi MH, Fava M, Rush AJ, Wisniewski S, Weissman MM. Children of depressed mothers 1 year after the initiation of maternal treatment: findings from the STAR*D-Child Study. Am J Psychiatry. 2008 Sep;165(9):1136-47. doi: 10.1176/appi.ajp.2008.07081286. Epub 2008 Jun 16. PMID 18558646
- [Background] Youth Risk Behavior Survey-Data Summary & Trends Report: 2007-2017. (2020). 91.
- [Background] Giano Z, Wheeler DL, Hubach RD. The frequencies and disparities of adverse childhood experiences in the U.S. BMC Public Health. 2020 Sep 10;20(1):1327. doi: 10.1186/s12889-020-09411-z. PMID 32907569
- [Background] Cook BL, McGuire T, Miranda J. Measuring trends in mental health care disparities, 2000 2004. Psychiatr Serv. 2007 Dec;58(12):1533-40. doi: 10.1176/ps.2007.58.12.1533. PMID 18048553
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Miles JN, Marshall GN, Schell TL. Spanish and English versions of the PTSD Checklist-Civilian version (PCL-C): testing for differential item functioning. J Trauma Stress. 2008 Aug;21(4):369-76. doi: 10.1002/jts.20349. PMID 18720394
- [Background] Haskett ME, Ahern LS, Ward CS, Allaire JC. Factor structure and validity of the parenting stress index-short form. J Clin Child Adolesc Psychol. 2006 Jun;35(2):302-12. doi: 10.1207/s15374424jccp3502_14. PMID 16597226